CLINICAL TRIAL: NCT01044134
Title: A 6-Month Study on Diet and Weight Loss in Overweight Adolescents
Brief Title: Think AHEAD (A Healthy Eating And Drinking) Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We achieved n=38, due to slow recruitment (=2/3 of target).
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, David S. Ludwig, MD, PhD, Professor, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: X09-11-0587
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet + Water (Experimental): Participants will be counseled to follow a standard weight-reducing diet including consumption of 1) ample vegetables, fruits, and legumes; 2) whole rather than refined grains; and 3) high-quality proteins at most meals and snacks. Moreover, we will recommend limiting intake of added fats and sugars and avoiding juices and sugar-sweetened beverages (per standard practice). Participants will also be counseled to increase their water intake to 8 cups per day, consistent with the popular "8 × 8" recommendation (eight 8-oz glasses of water).
  Interventions: Behavioral: Dietary counseling
- Diet (Active Comparator): Participants will be counseled on the same standard weight-reducing diet, as described above, with no specific advice regarding water consumption. Furthermore, no specific dietary recommendations will be provided on altering fluid/beverage intake, other than to decrease calorie-containing beverages as noted above. When participants ask for a recommendation regarding water intake, they will be advised that drinking plain water is the best way to satisfy thirst and instructed to drink when thirsty.
  Interventions: Behavioral: Dietary counseling

INTERVENTIONS:
Behavioral: Dietary counseling — Participants will receive personalized dietary counseling to promote behavior change

SUMMARY:
Advice to increase water consumption as part of a weight-reducing diet - typically to 8 cups (64 fl oz, ~2 L) per day ("8x8" water recommendation) - is almost ubiquitously recommended by healthcare professionals. Many believe that water promotes weight loss through numerous physiological mechanisms. However, only limited observational data and virtually no experimental data exist regarding the effects of water consumption on body weight. In this study, we propose a randomized controlled pilot study in which two groups of overweight adolescents will receive a standard weight loss regimen, either with (experimental intervention) or without (control intervention) additional advice and support to increase water consumption. We will utilize individual sessions, an innovative text messaging protocol, and motivational telephone calls to promote adherence to the interventions. The purpose of this pilot study is to evaluate feasibility and obtain preliminary efficacy data, to inform design of a future, definitive study.

It is hypothesized that increasing water consumption will improve the efficacy of a standard weight-reducing diet and will lead to decreased consumption of energy-containing beverages, decreased total energy intake, improved diet quality, improved immune status, and improved cardiovascular and diabetes risk factors. This simple behavioral intervention will be feasible and will significantly increase water consumption among participants in the experimental vs. control group.

DETAILED DESCRIPTION:
This is a 6-month randomized controlled trial. After the initial baseline screening and assessments, 60 overweight adolescents will be randomly assigned (30 subjects per group) to a standard weight-reducing diet with the advice to consume 8 cups of water per day (experimental group) or the same standard weight-reducing diet without additional advice (control group). The interventions will consist of nutrition education and behavioral counseling by a registered dietitian, during individual sessions and telephone calls. Mobile text messaging will be used to reinforce information presented at the individual sessions and thereby foster adherence to dietary advice. Diet prescriptions will differ only in regard to the specificity of recommendations regarding water consumption and physical activity recommendations will not differ between groups. The frequency and content of text messages will be consistent between the experimental and control groups, with the exception that the experimental group will receive an additional phrase with each message to encourage the "8 x8" water recommendation.

A registered dietitian will communicate with each participant one time per month, either during an individual session or by telephone. Individual sessions will include nutrition classes, taste testing, hands-on activities, and opportunities for questions and answers. Text messages will be sent on a daily basis.

Study outcomes will be assessed at baseline and at regular intervals throughout the 6 months of the study.

ANALYSIS PLAN:

The blinding of the randomization will be broken on or after July 28, 2014 and the data will be analyzed according to the following plan. All analyses will follow the intention-to-treat principle, attributing each subject to his or her assigned diet regardless of compliance. Baseline characteristics will be compared between the diet groups using the Fisher exact test for categorical variables and t-test for continuous variables. The 6-month change from baseline in the primary and secondary outcomes will be compared between groups using a general linear model, adjusting for baseline covariates that are potentially correlated with the outcome. These include demographics, socioeconomic status, anthropometrics, physical activity, and beverage consumption. We will further test covariates for potential interaction, i.e., differential effect on outcome in the two trial arms. The null hypothesis is that the 6-month change from baseline will not differ between diet groups.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 85th percentile for sex and age according to CDC growth charts
* Access to a working telephone and cell phone
* At least one parent willing and able to participate in the intervention with the subject
* Residing in predominately one household (no more than one weekend every two weeks in a secondary household)
* Medical clearance from a primary care provider or treating physician to rule out any major medical illness, disability, or disorder (e.g., liver disease, renal failure, cancer)

Exclusion Criteria:

* Intake of more than 4 cups (250 mL per cup) of water per day
* BMI ≥ 40 kg/m2
* Currently smoking (> 1 cigarette in the past week)
* Major surgery within the previous 6 months
* Does not have a primary care provider
* Physician diagnosis of a major medical illness (e.g. diabetes)
* Previous diagnosis of an eating disorder
* Physical, mental, or cognitive handicaps that prevent participation
* Chronic use of medications that may affect study outcomes (e.g. stimulants or diuretics)
* Another member of the family (first degree relative) or household participating in the study
* A friend, classmate or coworker participating in the study with whom they have contact with one or more times per week
* Girls who are pregnant, planning to become pregnant in the next 6 months, lactating, or within 6 months postpartum

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2011-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Body mass index | 6 month change

SECONDARY OUTCOMES:
Body fat percentage | 6 month change
Body circumferences | 6 month change
Urine specific gravity | Change throughout 6 months
Hunger, satiety, and palatability ratings | 6 month change
Diet quality | 6 month change
Satisfaction rating | 6 months
Immune status | 6 month change
Cardiovascular risk factors | 6 month change
Diabetes risk factors | 6 month change

CONTACTS AND LOCATIONS:
Overall Officials: David S Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Wong JMW, Ebbeling CB, Robinson L, Feldman HA, Ludwig DS. Effects of Advice to Drink 8 Cups of Water per Day in Adolescents With Overweight or Obesity: A Randomized Clinical Trial. JAMA Pediatr. 2017 May 1;171(5):e170012. doi: 10.1001/jamapediatrics.2017.0012. Epub 2017 May 1. PMID 28264082